CLINICAL TRIAL: NCT05553522
Title: Phase 1 Trial of Tucatinib, Trastuzumab, and Capecitabine With Stereotactic Radiosurgery (SRS) in Patients With Brain Metastases From HER-2 Positive Breast Cancer
Brief Title: Tucatinib, Trastuzumab, and Capecitabine With SRS for Brain Metastases From HER-2 Positive Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Baptist Health South Florida (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-AHL-001
Record Dates: First submitted 2022-09-16; First posted 2022-09-23 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2024-12

CONDITIONS: Brain Metastases; HER2-positive Breast Cancer
Keywords: brain metastases; HER2-positive breast cancer
MeSH Terms: conditions — Brain Neoplasms | interventions — tucatinib; Trastuzumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Investigational Treatment (Experimental)
  Interventions: Combination Product: Combined use of SRS with Tucatinib, Trastuzumab, and Capecitabine

INTERVENTIONS:
Combination Product: Combined use of SRS with Tucatinib, Trastuzumab, and Capecitabine — SRS and oral tucatinib for 2 wk, followed by oral tucatinib, oral capecitabine, and intravenous (IV) trastuzumab maintenance during 21-d cycles until tumor progression, participant withdrawal, a severe adverse event deemed related to the study drug, or the treating physician discontinues the drug. There are three dosing levels of tucatinib (Dose Level 0, Dose Level -1, or Dose Level -2) using a dose de-escalation scheme. Dosing of capectabine (1000 mg/m2 BID Days 1-14) and trastuzumab (6 mg/kg once per 21 days; 8 mg/kg initial loading dose) per cycle will remain the same regardless of tucatinib dosing.
  Dose Level 0: 300 mg twice a day (BID) continuously for 2 wk post SRS, then 300 mg BID continuously per cycle.
  Dose Level -1: 250 mg twice a day (BID) continuously for 2 wk post SRS, then 250 mg BID continuously per cycle.
  Dose Level -2: 200 mg twice a day (BID) continuously for 2 wk post SRS, then 200 mg BID continuously per cycle.

SUMMARY:
This research study will evaluate how well brain metastases associated with HER-2 positive breast cancer can be controlled using a type of radiation known as stereotactic radiosurgery (SRS) when combined with three therapeutic agents, tucatinib, capecitabine, and trastuzumab.

The combined use of SRS with the three drugs is considered investigational.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed HER-2 -positive breast cancer with newly-diagnosed brain metastases.
2. ECOG Performance Status (PS) of 0, 1, 2
3. Patients with 1-10 brain metastases will be candidates for tucatinib, capecitabine, and trastuzumab with SRS at the discretion of the treating radiation oncologist. Intra-cranial brain metastasis must measure 3 cm or less in the greatest dimension
4. Age 18 years or greater and being willing and able to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures
5. Life expectancy at least 12 weeks
6. Any number of prior systemic therapies will be allowed, except tucatinib and capecitabine.
7. Hemoglobin ≥ 9g/dL, White blood count ≥3.0 × 10^9/ L , Absolute Granulocyte count ≥1.5x 10^9/ L and platelet count ≥100 × 10^9/ L.
8. Serum bilirubin ≤ 1.5 × ULN
9. AST and / or ALT <= 2 × ULN (≤ 5 × ULN when clearly attributable to the presence of liver metastases)
10. Serum creatinine ≤ 1.5 × ULN or calculated creatinine clearance > 60mL/min
11. Ability to comply with study procedures and monitoring
12. For women of childbearing potential, a negative pregnancy test should be obtained within one week prior to the start of therapy
13. Male or female patients of reproductive potential need to employ two highly effective and acceptable forms of contraception throughout their participation in the study and for 7 months after last dose of tucatinib, capecitabine and trastuzumab.

Highly effective and acceptable forms of contraception are:

* Male condom plus spermicide
* Cap plus spermicide
* Diaphragm plus spermicide
* Copper T
* Progesterone T
* Levonorgestrel-releasing intrauterine system (e.g., Mirena®)
* Implants
* Hormone shot or injection
* Combined pill
* Mini-pill
* Patch

Postmenopausal woman on the study (that will not need contraception) is defined as:

* Amenorrhoeic for 1 year or more following cessation of exogenous hormonal treatments
* LH and FSH levels in the postmenopausal range for women under 50
* Radiation-induced oophorectomy with last menses > 1 year ago
* Chemotherapy-induced menopause with >1 year interval since last menses
* Surgical sterilization (bilateral oophorectomy or hysterectomy).

Men and women and members of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

1. Patients with leptomeningeal metastases documented by MRI or CSF evaluation
2. Evidence of intra-tumoral or peri-tumoral hemorrhage deemed significant by the treating physician
3. Brain metastases within 5 mm of the optic chiasm or optic nerve
4. Significant or recent acute gastrointestinal disorders with diarrhea as a major symptom, e.g., Crohn's disease, malabsorption, or CTCAE grade >2 diarrhea of any etiology at baseline
5. History of clinically significant or uncontrolled cardiac disease, including congestive heart failure, angina, myocardial infarction, arrhythmia, New York Heart Association (NYHA) functional classification of 3 or 4
6. Unable to undergo brain MRI
7. Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C
8. All toxicities from prior therapies must have resolved to CTCAE v 5.0 grade 1 or better by the time of study enrollment
9. Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., active or uncontrolled infection, uncontrolled diabetes, second active malignancy) that could cause unacceptable safety risks or compromise compliance with the protocol
10. Currently receiving other investigational cancer therapy within 4 weeks prior to start of study treatment with the exception of continuing therapy with GnRH analogues
11. Mean QT interval corrected heart rate (QTc) ≥ 470ms calculated from 3 electrocardiograms using Frediricia's Correction
12. Left ventricular ejection fraction (LVEF) <50%
13. Concomitant use of strong cytochrome P450 (CYP)3A inhibitors including macrolide antibiotics (e.g., Telithromycin), antifungals (e.g., Itraconazole), antivirals (e.g., ritonavir), and Nefazodone
14. Concomitant use of strong CYP2C8 inhibitor within 5 half-lives of the inhibitor
15. Concomitant use of strong CYP3A4 inducers (e.g., phenytoin, rifampicin, carbamazepine, St. John's Wort) within 5 days prior to the first dose of study treatment
16. Concomitant use of a strong CYP2C8 inducer within 5 days prior to the first dose of study treatment
17. History of hypersensitivity to tucatinib, capecitabine, and trastuzumab, or any of its excipients
18. History and/or confirmed corneal ulceration
19. Pregnant or breast feeding
20. Use of anthracyline will be prohibited on the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | During first 4 weeks following SRS
  Toxicities will be graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0). DLTs are defined as any of the following events:
  1. Grade 3 or 4 thrombocytopenia
  2. Grade 4 anemia
  3. Grade 4 neutropenia lasting more than 7 days
  4. Febrile neutropenia
  5. Any non-hematologic toxicity of grade 3 or greater (excluding alopecia) despite maximal medical therapy
  6. Grade 4 radiation-induced skin changes
  7. Any episode of noninfectious pneumonitis.
Incidence of radiation-related toxicities | 30 days of progression or last dose of drug
  Toxicities presumed to be due to radiation are defined as:
  1. Acute, < 90 days from treatment start: Expected toxicities include hair loss (for lesions abutting skull), erythema of the scalp (for lesions abutting skull), headache, nausea, and vomiting. Reactions in the ear canals and on the ear should be observed and treated symptomatically. Pin site infection, pin site pain, facial swelling/bruising, and scalp numbness are other common acute effects. Acute toxicity is defined by CTCAE v5.0.
  2. Both acute and delayed, > or = 90 days from treatment start (lethargy, transient worsening of existing neurological deficits) or late (radiation necrosis, cognitive dysfunction, accelerated atherosclerosis, radiation-induced neoplasms) effects of radiotherapy are to be recorded and included in the toxicity evaluation. Late or delayed toxicity is defined by CTCAE v5.0.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Six months
  Time from first dose of study drug until the first date of disease progression or death due any cause. The date of disease progression will be defined as the earliest date of disease progression based on central review. For participants whose disease has not progressed at the time of the analysis, censoring will be performed using the date of the last valid disease assessment. The data will be analyzed by the Kaplan-Meier method. PFS will be considered when there is progression just intracranially, as well as when there is progression intracranially or extracranially.
Overall survival | One year
  Time from the beginning of study drug treatment until death due to any cause. For participants who have not died at the time of the analysis, censoring will be performed using the date the patient was last known to be alive. The data will be analyzed by the Kaplan-Meier method.
Overall response rate (ORR) | One year
  Proportion of participants with a complete response (CR) or partial response (PR) as defined by Response Evaluation Criteria in Solid Tumours (RECIST) 1.1. For ORR analysis in all the treated population, participants with an CR or PR will be counted as successes and all other participants (including those with missing response information) will be counted as failures. ORR will be considered for intracranial and extracranial tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Manmeet Ahluwalia, M.D., MBA, Principal Investigator — Miami Cancer Institute/Baptist Health South Florida
Locations (1):
- Miami Cancer Institute at Baptist Health, Inc., Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ahluwalia MS, Vogelbaum MV, Chao ST, Mehta MM. Brain metastasis and treatment. F1000Prime Rep. 2014 Dec 1;6:114. doi: 10.12703/P6-114. eCollection 2014. PMID 25580268
- [Background] Moulder SL, Borges VF, Baetz T, Mcspadden T, Fernetich G, Murthy RK, Chavira R, Guthrie K, Barrett E, Chia SK. Phase I Study of ONT-380, a HER2 Inhibitor, in Patients with HER2+-Advanced Solid Tumors, with an Expansion Cohort in HER2+ Metastatic Breast Cancer (MBC). Clin Cancer Res. 2017 Jul 15;23(14):3529-3536. doi: 10.1158/1078-0432.CCR-16-1496. Epub 2017 Jan 4. PMID 28053022
- [Background] Morikawa A, Peereboom DM, Thorsheim HR, Samala R, Balyan R, Murphy CG, Lockman PR, Simmons A, Weil RJ, Tabar V, Steeg PS, Smith QR, Seidman AD. Capecitabine and lapatinib uptake in surgically resected brain metastases from metastatic breast cancer patients: a prospective study. Neuro Oncol. 2015 Feb;17(2):289-95. doi: 10.1093/neuonc/nou141. Epub 2014 Jul 11. PMID 25015089
- [Background] Geyer CE, Forster J, Lindquist D, Chan S, Romieu CG, Pienkowski T, Jagiello-Gruszfeld A, Crown J, Chan A, Kaufman B, Skarlos D, Campone M, Davidson N, Berger M, Oliva C, Rubin SD, Stein S, Cameron D. Lapatinib plus capecitabine for HER2-positive advanced breast cancer. N Engl J Med. 2006 Dec 28;355(26):2733-43. doi: 10.1056/NEJMoa064320. PMID 17192538
- [Background] Pheneger T, Bouhana K, Anderson D, Garrus J, Ahrendt K, Allen S, et al. In Vitro and in vivo activity of ARRY-380: A potent, small molecule inhibitor of ErbB2. AACR Annual Meeting-- Apr 18-22, 2009; Denver, CO. Abstract #1795.
- [Background] Murthy R, Borges VF, Conlin A, Chaves J, Chamberlain M, Gray T, Vo A, Hamilton E. Tucatinib with capecitabine and trastuzumab in advanced HER2-positive metastatic breast cancer with and without brain metastases: a non-randomised, open-label, phase 1b study. Lancet Oncol. 2018 Jul;19(7):880-888. doi: 10.1016/S1470-2045(18)30256-0. Epub 2018 May 24. PMID 29804905
- [Background] Lin NU, Borges V, Anders C, Murthy RK, Paplomata E, Hamilton E, Hurvitz S, Loi S, Okines A, Abramson V, Bedard PL, Oliveira M, Mueller V, Zelnak A, DiGiovanna MP, Bachelot T, Chien AJ, O'Regan R, Wardley A, Conlin A, Cameron D, Carey L, Curigliano G, Gelmon K, Loibl S, Mayor J, McGoldrick S, An X, Winer EP. Intracranial Efficacy and Survival With Tucatinib Plus Trastuzumab and Capecitabine for Previously Treated HER2-Positive Breast Cancer With Brain Metastases in the HER2CLIMB Trial. J Clin Oncol. 2020 Aug 10;38(23):2610-2619. doi: 10.1200/JCO.20.00775. Epub 2020 May 29. PMID 32468955
- [Background] Brown PD, Jaeckle K, Ballman KV, Farace E, Cerhan JH, Anderson SK, Carrero XW, Barker FG 2nd, Deming R, Burri SH, Menard C, Chung C, Stieber VW, Pollock BE, Galanis E, Buckner JC, Asher AL. Effect of Radiosurgery Alone vs Radiosurgery With Whole Brain Radiation Therapy on Cognitive Function in Patients With 1 to 3 Brain Metastases: A Randomized Clinical Trial. JAMA. 2016 Jul 26;316(4):401-409. doi: 10.1001/jama.2016.9839. PMID 27458945
- [Background] Slamon DJ, Clark GM, Wong SG, Levin WJ, Ullrich A, McGuire WL. Human breast cancer: correlation of relapse and survival with amplification of the HER-2/neu oncogene. Science. 1987 Jan 9;235(4785):177-82. doi: 10.1126/science.3798106.
- [Background] Aragon-Ching JB, Zujewski JA. CNS metastasis: an old problem in a new guise. Clin Cancer Res. 2007 Mar 15;13(6):1644-7. doi: 10.1158/1078-0432.CCR-07-0096. PMID 17363516
- [Background] Sperduto PW, Kased N, Roberge D, Xu Z, Shanley R, Luo X, Sneed PK, Chao ST, Weil RJ, Suh J, Bhatt A, Jensen AW, Brown PD, Shih HA, Kirkpatrick J, Gaspar LE, Fiveash JB, Chiang V, Knisely JP, Sperduto CM, Lin N, Mehta M. Summary report on the graded prognostic assessment: an accurate and facile diagnosis-specific tool to estimate survival for patients with brain metastases. J Clin Oncol. 2012 Feb 1;30(4):419-25. doi: 10.1200/JCO.2011.38.0527. Epub 2011 Dec 27. PMID 22203767
- [Background] Brufsky AM, Mayer M, Rugo HS, Kaufman PA, Tan-Chiu E, Tripathy D, Tudor IC, Wang LI, Brammer MG, Shing M, Yood MU, Yardley DA. Central nervous system metastases in patients with HER2-positive metastatic breast cancer: incidence, treatment, and survival in patients from registHER. Clin Cancer Res. 2011 Jul 15;17(14):4834-43. doi: 10.1158/1078-0432.CCR-10-2962. PMID 21768129
- [Background] Romond EH, Perez EA, Bryant J, Suman VJ, Geyer CE Jr, Davidson NE, Tan-Chiu E, Martino S, Paik S, Kaufman PA, Swain SM, Pisansky TM, Fehrenbacher L, Kutteh LA, Vogel VG, Visscher DW, Yothers G, Jenkins RB, Brown AM, Dakhil SR, Mamounas EP, Lingle WL, Klein PM, Ingle JN, Wolmark N. Trastuzumab plus adjuvant chemotherapy for operable HER2-positive breast cancer. N Engl J Med. 2005 Oct 20;353(16):1673-84. doi: 10.1056/NEJMoa052122. PMID 16236738
- [Background] Baselga J, Cortes J, Kim SB, Im SA, Hegg R, Im YH, Roman L, Pedrini JL, Pienkowski T, Knott A, Clark E, Benyunes MC, Ross G, Swain SM; CLEOPATRA Study Group. Pertuzumab plus trastuzumab plus docetaxel for metastatic breast cancer. N Engl J Med. 2012 Jan 12;366(2):109-19. doi: 10.1056/NEJMoa1113216. Epub 2011 Dec 7. PMID 22149875
- [Background] Pestalozzi BC, Brignoli S. Trastuzumab in CSF. J Clin Oncol. 2000 Jun;18(11):2349-51. doi: 10.1200/JCO.2000.18.11.2349. No abstract available. PMID 10829059
- [Background] Rusnak DW, Lackey K, Affleck K, Wood ER, Alligood KJ, Rhodes N, Keith BR, Murray DM, Knight WB, Mullin RJ, Gilmer TM. The effects of the novel, reversible epidermal growth factor receptor/ErbB-2 tyrosine kinase inhibitor, GW2016, on the growth of human normal and tumor-derived cell lines in vitro and in vivo. Mol Cancer Ther. 2001 Dec;1(2):85-94. PMID 12467226
- [Background] Leone JP, Lee AV, Brufsky AM. Prognostic factors and survival of patients with brain metastasis from breast cancer who underwent craniotomy. Cancer Med. 2015 Jul;4(7):989-94. doi: 10.1002/cam4.439. Epub 2015 Mar 9. PMID 25756607
- See also: FDA Drugs development approval process — https://www.fda.gov/Drugs/DevelopmentApprovalProcess/DevelopmentResources/DrugInteractionsLabeling/ucm093664.htm#table3-1)
- See also: Miami Cancer Institute — https://cancer.baptisthealth.net/